CLINICAL TRIAL: NCT02383212
Title: A First-in-Human Study of Repeat Dosing With REGN2810, a Monoclonal, Fully Human Antibody to Programmed Death - 1 (PD-1), as Single Therapy and in Combination With Other Anti-Cancer Therapies in Patients With Advanced Malignancies
Brief Title: Study of REGN2810 (Anti-PD-1) in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R2810-ONC-1423; 2015-002132-41 (EudraCT Number)
Record Dates: First submitted 2015-02-02; First posted 2015-03-09 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Advanced Cancer; Advanced Malignancies
Keywords: Advanced cancerous growth
MeSH Terms: interventions — cemiplimab; Radiation Dose Hypofractionation; Cyclophosphamide; Docetaxel; Carboplatin; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim; Paclitaxel; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Monotherapy Cohort (Experimental): Cemiplimab will be administered alone
  Interventions: Drug: Cemiplimab
- Dual Combination Cohorts (Experimental): Doses of cemiplimab will be administered in combination with hypofractionated radiotherapy
  Doses of cemiplimab will be administered in combination with Cyclophosphamide
  Doses of cemiplimab will be administered in combination with Docetaxel
  Interventions: Drug: Cemiplimab; Radiation: Hypofractionated radiotherapy; Drug: Cyclophosphamide; Drug: Docetaxel
- Triple Combination Cohorts (Experimental): Doses of cemiplimab will be administered in combination with hypofractionated radiotherapy plus Cyclophosphamide
  Doses of cemiplimab will be administered in combination with hypofractionated radiotherapy plus GM-CSF
  Doses of cemiplimab will be administered in combination with Carboplatin plus Paclitaxel
  Doses of cemiplimab will be administered in combination with Carboplatin plus Pemetrexed
  Doses of cemiplimab will be administered in combination with Carboplatin plus Docetaxel
  Interventions: Drug: Cemiplimab; Radiation: Hypofractionated radiotherapy; Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Carboplatin; Drug: GM-CSF; Drug: Paclitaxel; Drug: Pemetrexed
- Quadruple Combination Cohorts (Experimental): Doses of cemiplimab will be administered in combination with hypofractionated radiotherapy plus GM-CSF plus Cyclophosphamide
  Interventions: Drug: Cemiplimab; Radiation: Hypofractionated radiotherapy; Drug: Cyclophosphamide; Drug: GM-CSF

INTERVENTIONS:
Drug: Cemiplimab
  Other Names: REGN2810; Libtayo
Radiation: Hypofractionated radiotherapy
  Arms: Dual Combination Cohorts; Quadruple Combination Cohorts; Triple Combination Cohorts
Drug: Cyclophosphamide
  Arms: Dual Combination Cohorts; Quadruple Combination Cohorts; Triple Combination Cohorts
Drug: Docetaxel
  Arms: Dual Combination Cohorts; Triple Combination Cohorts
Drug: Carboplatin
  Arms: Triple Combination Cohorts
Drug: GM-CSF
  Other Names: LEUKINE®
  Arms: Quadruple Combination Cohorts; Triple Combination Cohorts
Drug: Paclitaxel
  Arms: Triple Combination Cohorts
Drug: Pemetrexed
  Arms: Triple Combination Cohorts

SUMMARY:
This is a phase 1, open-label, multicenter, ascending-dose escalation study of cemiplimab, alone and in combination with other anti-cancer therapies in patients with advanced malignancies.

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of malignancy with demonstrated progression of a solid tumor (non-lymphoma) with no alternative standard-of-care therapeutic option (certain exceptions may apply).
2. At least 1 measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria for response assessment (certain exceptions may apply)
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Key Exclusion Criteria:

1. Ongoing or recent (within 5 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments, which may suggest risk for immune-related adverse events (irAEs). The following are not exclusionary: vitiligo, childhood asthma that has resolved, residual hypothyroidism that required only hormone replacement or psoriasis that does not require systemic treatment.
2. Prior treatment with an agent that blocks the programmed death-1/ programmed death-ligand 1 (PD-1/PD-L1 pathway) (certain exceptions may apply)
3. Prior treatment with other immune modulating agents within fewer than 4 weeks prior to the first dose of cemiplimab. Examples of immune modulating agents include blockers of CTLA-4, 4-1BB (CD137), OX-40, therapeutic vaccines, or cytokine treatments.
4. Untreated brain metastasis(es) that may be considered active. Patients with previously treated brain metastases may participate provided they are stable (i.e., without evidence of progression by imaging for at least 6 weeks prior to the first dose of study treatment, and any neurologic symptoms have returned to baseline), and there is no evidence of new or enlarging brain metastases, and the patient does not require any systemic corticosteroids for management of brain metastases within 4 weeks prior to the first dose of cemiplimab (certain exceptions may apply).
5. Immunosuppressive corticosteroid doses (>10 mg prednisone daily or equivalent) within 4 weeks prior to the first dose of cemiplimab

The information provided above is not intended to contain all considerations relevant to potential participation in a clinical trial, therefore not all inclusion/ exclusion criteria are listed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2015-02-02 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (TEAEs) | Change from baseline to week 48
  Primary safety variables include incidence and severity of TEAEs, abnormal laboratory findings and number of participants with dose limiting toxicities (DLTs)
Incidence of abnormal laboratory findings | Change from baseline to week 48
Number of participants with dose limiting toxicities (DLTs) | Change from baseline to 28 days after first dose of cemiplimab

SECONDARY OUTCOMES:
Response Evaluation Criteria in Solid Tumors (RECIST) as measured by Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) | Change from baseline to week 48
Immune-Related Response Criteria (irRC) applied to RECIST measurements | Change from baseline to week 48
Incidence of development of anti-cemiplimab antibodies | Up to week 48
Antitumor activity measured by progression-free survival (PFS) | Up to 72 weeks
Antitumor activity measured by overall survival | Up to 249 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (47):
- United States (40):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Western Regional Medical Center, Goodyear, Arizona
  - Mayo Clinic, Phoenix, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - City of Hope National Medical Center, Duarte, California
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Stanford University, Stanford, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Norwalk Hospital, Norwalk, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Cancer Center, Fairway, Kansas
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Center, Detroit, Michigan
  - Washington University School of Medicine Siteman Cancer Center, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Columbia University Medical Center, New York, New York
  - Laura & Isaac Perlmutter Cancer Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Duke Cancer Institute, Durham, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Medical Center Shadyside, Pittsburgh, Pennsylvania
  - Miriam Hospital, Providence, Rhode Island
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Mary Crowley Cancer Research Center - Medical City, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - START South Texas Accelerated Research Therapeutics, San Antonio, Texas
  - Northwest Medical Specialties, Tacoma, Washington
- Peter Maccallum Cancer Centre, Melbourne, Australia
- Spain (6):
  - Institut Catala d'Oncologia L'hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario HM Sanchinarro-CIOCC, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - MD Anderson Cancer Center, Madrid

REFERENCES:
- [Derived] Babiker H, Brana I, Mahadevan D, Owonikoko T, Calvo E, Rischin D, Moreno V, Papadopoulos KP, Crittenden M, Formenti S, Giralt J, Garrido P, Soria A, Hervas-Moron A, Mohan KK, Fury M, Lowy I, Mathias M, Feng M, Li J, Stankevich E. Phase I Trial of Cemiplimab, Radiotherapy, Cyclophosphamide, and Granulocyte Macrophage Colony-Stimulating Factor in Patients with Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma. Oncologist. 2021 Sep;26(9):e1508-e1513. doi: 10.1002/onco.13810. Epub 2021 May 22. PMID 33942954
- [Derived] Moreno V, Garrido P, Papadopoulos KP, De Miguel Luken MJ, Gil-Martin M, Aljumaily R, Rosen LS, Rietschel P, Mohan KK, Yoo SY, Stankevich E, Lowy I, Fury MG. Tolerability and antitumor activity of cemiplimab, a human monoclonal anti-PD-1, as monotherapy in patients with pretreated non-small cell lung cancer (NSCLC): Data from the Phase 1 NSCLC expansion cohort. Lung Cancer. 2021 May;155:151-155. doi: 10.1016/j.lungcan.2021.02.034. Epub 2021 Mar 4. PMID 33831732
- [Derived] Rischin D, Migden MR, Lim AM, Schmults CD, Khushalani NI, Hughes BGM, Schadendorf D, Dunn LA, Hernandez-Aya L, Chang ALS, Modi B, Hauschild A, Ulrich C, Eigentler T, Stein B, Pavlick AC, Geiger JL, Gutzmer R, Alam M, Okoye E, Mathias M, Jankovic V, Stankevich E, Booth J, Li S, Lowy I, Fury MG, Guminski A. Phase 2 study of cemiplimab in patients with metastatic cutaneous squamous cell carcinoma: primary analysis of fixed-dosing, long-term outcome of weight-based dosing. J Immunother Cancer. 2020 Jun;8(1):e000775. doi: 10.1136/jitc-2020-000775. PMID 32554615
- [Derived] Migden MR, Rischin D, Schmults CD, Guminski A, Hauschild A, Lewis KD, Chung CH, Hernandez-Aya L, Lim AM, Chang ALS, Rabinowits G, Thai AA, Dunn LA, Hughes BGM, Khushalani NI, Modi B, Schadendorf D, Gao B, Seebach F, Li S, Li J, Mathias M, Booth J, Mohan K, Stankevich E, Babiker HM, Brana I, Gil-Martin M, Homsi J, Johnson ML, Moreno V, Niu J, Owonikoko TK, Papadopoulos KP, Yancopoulos GD, Lowy I, Fury MG. PD-1 Blockade with Cemiplimab in Advanced Cutaneous Squamous-Cell Carcinoma. N Engl J Med. 2018 Jul 26;379(4):341-351. doi: 10.1056/NEJMoa1805131. Epub 2018 Jun 4. PMID 29863979
- [Derived] Falchook GS, Leidner R, Stankevich E, Piening B, Bifulco C, Lowy I, Fury MG. Responses of metastatic basal cell and cutaneous squamous cell carcinomas to anti-PD1 monoclonal antibody REGN2810. J Immunother Cancer. 2016 Nov 15;4:70. doi: 10.1186/s40425-016-0176-3. eCollection 2016. PMID 27879972